CLINICAL TRIAL: NCT01389440
Title: Phase II Study Open, Not Randomized to Evaluate the Efficacy and Safety of Neoadjuvant Treatment With Gemcitabine and Erlotinib Followed by Gemcitabine, Erlotinib and Radiotherapy in Patients With Resectable Pancreatic Adenocarcinoma
Brief Title: Efficacy and Safety of a Neoadjuvant Treatment in Pancreatic Cancer
Acronym: GEMCAD1003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD1003; 2010-021738-72 (EudraCT Number)
Record Dates: First submitted 2011-07-01; First posted 2011-07-08 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Resectable pancreatic adenocarcinoma; Gemcitabine; Erlotinib; Radiotherapy; Neoadjuvant treatment
MeSH Terms: interventions — Gemcitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, Erlotinib and radiotherapy (Experimental): Gemcitabine + Erlotinib follow by Gemcitabine + Erlotinib + radiotherapy
  Interventions: Drug: Gemcitabine and Erlotinib

INTERVENTIONS:
Drug: Gemcitabine and Erlotinib — Administration of gemcitabine (300mg/m2/weekly)with Erlotinib (100 mg/daily) and radiotherapy (45 Gy/daily) after a period of infusion with a full dose of Gemcitabine (1.000mg/m2/weekly) and Erlotinib (100 mg/daily)
  Other Names: Gemcitabine and Tarceva

SUMMARY:
This is a Phase II open study, not randomized with a neoadjuvant therapy,combination of Gemcitabine (1,000 mg/m2/week) with Erlotinib (100mg/day) (3 cycles of 4 weeks), followed by gemcitabine (300 mg/m2/week) combined with Erlotinib (100mg/day) and radiotherapy (45 Gy / day fr180 cGy) (5 cycles of 1 week) in patients with resectable pancreatic adenocarcinoma to assess the percentage of R0 resections. They have planned a total of 21 visits.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign the inform consent form
* Age between 18-75 years
* Subject has not undergone any chemotherapy or radiotherapy previously
* Functional status o-1 (ECOG scale)
* Satisfy all radiological inclusion criteria (MSCT performed 28 days before the treatment starts and a centralized evaluation)
* Patients with a cytologically confirmed diagnosis of pancreatic adenocarcinoma(preferably by EUS)
* Appropriate analytical as inclusion criteria (7 days before the treatment starts):
* bone marrow status: neutrophils ≥ 1,500x10^9/L; platelets ≥ 100x10^9/L; hemoglobin ≥ 9g/dL.
* INR ≤ 1.5 and PTT ≤ 1.5 x upper range of normal.
* Bilirubin ≤ 5 mg/dL
* Albumin> 34 g/L
* Renal function: creatinine ≤ 1.5 mg/dL and creatinine clearance> 50ml/min

Exclusion Criteria:

* patients treated with any of the study's drugs
* patients who has develop other primary tumors in 5 years prior to the inclusion at the clinical trial, except for cervix carcinoma in situ or basal cell skin cancer which have been treated properly.
* significant clinical cardiovascular disease: stroke (≤ 6 months before the study inclusion), heart attack (≤ 6 months before inclusion), unstable ango pectoris, congestive heart failure second grade or higher of the New York Heart Association (NYHA) or serious cardiac arrhythmia requiring medication, uncontrolled hypertension
* Total o partial bowel obstruction
* Chronic diarrhea
* Current treatment with another investigational drug or participation in another clinical trial within 30 days prior to inclusion.
* Known hypersensitivity to any of the study drugs or their components
* Currently o recent therapeutic treatment (opposite to prophylactic) with oral or parenteral anticoagulants (full dose) or thrombolytic agents. Patients who receive (or are candidates to receive) anticoagulants for prophylaxis of cardiovascular risk, should continue (or begin) treatment at baseline
* Thromboembolic event history or bleeding in the 6 months prior to treatment.
* Evidence of bleeding diathesis or coagulopathy.
* Serious problems in wounds healing, ulcers or bone fractures.
* Major surgery, open biopsy or significant traumatic injury 28 days before treatment.
* Any other disease, metabolic disorder, physical examination findings or clinical laboratory that provides reasonable evidence for suspecting a disease or condition for which it is contraindicated or patient an experimental drug at high risk of experiencing complications related to treatment .
* Patients undergoing with organ allografts requiring immunosuppressive treatment.
* Pregnant or breastfeeding woman. It requires a negative pregnancy test (serum or urine) within 7 days before previous to treatment.
* Men and women of childbearing potential (including women who have had their last menstrual period in less than 2 years) not using effective contraception precautions
* Positive HIV status
* Addiction to alcohol or other drugs
* Known liver cirrhosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2016-11 (Actual); Study Completion 2017-01-22 (Actual)

PRIMARY OUTCOMES:
Percentage of ancients undergoing with neoadjuvant chemoradiotherapy and R0 resection | 3 years

SECONDARY OUTCOMES:
To describe the safety of the treatment | 3 years
  Based in safety population, all safety parameters will be analyzed and they will be recorded in lists and spread sheets. Most extreme intensity will be used for the notification of adverse events.
  Safety population will include all subjects that have taken at least one study medication dose.
Evaluate the response rate using RECIST criteria | 3 years
Evaluate the percentage of resectability | 3 years
Evaluate the percentage of lymphatic nodes removed | 3 years
Evaluate the percentage of lymphatic nodes involved | 3 years
Evaluate the pathological regression stage (primary tumor and lymphatic nodes) | 3 years
Relate RECIST criteria with the pathological regress stage | 3 years
Measure the progression free survival (time from the inclusion date to the progression of the disease or death) | 3 years
Evaluate the overall survival time | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Joan Maurel, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (10):
- Spain (10):
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
  - Institut Català d'Oncologia (ICO) de L'Hospitalet, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Santa Creu y Sant Pau, Hospital Sant Pau, Barcelona
  - Instituto Catalán de Oncología, Girona
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital la Fe de Valencia, Valencia
  - Clínico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Maurel J, Sanchez-Cabus S, Laquente B, Gaba L, Visa L, Fabregat J, Poves I, Rosello S, Diaz-Beveridge R, Martin-Richard M, Rodriguez J, Sabater L, Conill C, Cambray M, Reig A, Ayuso JR, Valls C, Ferrandez A, Bombi JA, Gines A, Garcia-Albeniz X, Fernandez-Cruz L. Outcomes after neoadjuvant treatment with gemcitabine and erlotinib followed by gemcitabine-erlotinib and radiotherapy for resectable pancreatic cancer (GEMCAD 10-03 trial). Cancer Chemother Pharmacol. 2018 Dec;82(6):935-943. doi: 10.1007/s00280-018-3682-9. Epub 2018 Sep 17. PMID 30225601